CLINICAL TRIAL: NCT04990518
Title: Physical Deconditioning and Non-Specific Low Back Pain: the PHYDEL Study. A Prospective Study in a COVID-19 Positive Cohort
Brief Title: Physical Deconditioning in COVID-19 Positive Patients and Non-Specific Low Back Pain
Acronym: Phydel
Status: Terminated | Type: Observational
Why Stopped: Grant not allowed
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Stephane Genevay, Principal investigator, University Hospital, Geneva
Other Study IDs: 2020-01994
Record Dates: First submitted 2021-07-22; First posted 2021-08-04 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Low Back Pain, Mechanical
Keywords: Low back pain; Physical deconditioning; Chronicity
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to take advantage of cohorts of patients followed for Coronavirus Disease 2019 (COVID19) expected to present poor physical fitness as the consequence of COVID19 to explore the relationship between physical fitness and low back pain (LBP). Level of physical fitness will be measured at baseline and incidence and intensity of LBP will be recoreded over 1 year.

DETAILED DESCRIPTION:
Non-specific low back pain (LBP) is the worldwide number one cause for disease related years lived with disability. It is frequently assumed that a low physical fitness is a major risk factor for acute LBP as well as a factor for chronic LBP. However only few prospective observational study have been conducted.

The purpose of this study is to take advantage of cohorts of patients followed for Coronavirus Disease 2019 (COVID19) expected to present poor physical fitness as the consequence of COVID19 and assessing level of physical fitness and both incidence and intensity of LBP over a 1-year period.

The study aims to determine if a poor physical health, as measured by 6 minutes walk test (6MWT) and 30''seconds sit to stand test (30''STS), is a risk factor for LBP occurrence and for chronic LBP Secondary objectives aim to explore the respective weight of physical factors (i.e. physical fitness, BMI, smoking, physical activities) and psychological factors (i.e. depression, anxiety, catastrophism, fear-avoidance) on the occurrence and severity of LBP.

According to the literature, we expect that in the physically healthy population, 15% will developed back pain; whereas in the population in poor physical health the incidence at 1 year will be 30%. If alpha error is set at 0.05 then 236 patients are required to have a 80% chance to confirm our hypothesis. In order to account for drop out, and considering that the risk of drop out is high in this type of non-interventional study 350 persons will be recruited. Note that this amount of persons should yield approximately 70 persons with low back pain, which allow up to 7 independent variable in a logistic or cox regression. This is based on the rule of at least 10 events (low back pain) per variable.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years, <65 years old
* Confirmed or supected COVID19 test
* Informed Consent as documented by signature

Exclusion Criteria:

* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant.
* Previous enrolment into the current study.
* Any comorbidity which could impact on the physical test (6-minutes walking test), e.g hip or knee osteoarthritis, polyneuropathy, symptomatic coronary heart disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People with a positive COVID test during the previous year, living in Geneva Switzerland, who declare their willingness to participate in clinical studies.
Sampling Method: Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2022-11-05 (Actual); Primary Completion 2022-11-05 (Actual); Study Completion 2022-11-05 (Actual)

PRIMARY OUTCOMES:
1-year incidence of LBP | 1 year
  Influence of baseline physical fitness on the number of participant with at least 1 episode of Low Back Pain
1-year incidence of chronic LBP | 1 year
  Influence of baseline physical fitness on the number of participant with at least 3 months of LBP most of the days

SECONDARY OUTCOMES:
Severity of LBP according to Pain trajectories | at least 3 months during the last year
  Influence of baseline physical fitness on 1 year pain trajectories recorded at the end of the study
Severity of LBP according to multiaxial evaluation | 1 year
  Influence of baseline physical fitness on Severity measured with COMI, multi-axial PRO specific for LBP
Severity of LBP according to treatment use | 1 year
  Influence of baseline physical fitness on the number of medical and paramedical appointements during the pain period
Influence of depression on 1-year incidence of LBP | 1 year
  Influence of depression as measured with HADS on the incidence of LBP
Influence of anxiety on 1-year incidence of LBP | 1 year
  Influence of anxiety as measured with HADS on the incidence of LBP
Influence of catastrophism on 1-year incidence of LBP | 1 year
  Influence of catastrpphism as measured with PCS on the incidence of LBP
Influence of fear-avoidance beliefs on 1-year incidence of LBP | 1 year
  Influence of fear-avoidance beliefs as measured with FABQ on the incidence of LBP
Influence of self-efficacy on 1-year incidence of LBP | 1 year
  Influence of self-efficacy as measured with PSEQ-2 on the incidence of LBP
Influence of depression on 1-year incidence of chronic LBP | 1 year
  Influence of depression as measured with HADS on the incidence of people with LBP for more than 3 months
Influence of anxiety on 1-year incidence of chronic LBP | 1 year
  Influence of anxiety as measured with HADS on the incidence of people with LBP for more than 3 months
Influence of catastrophism on 1-year incidence of chronic LBP | 1 year
  Influence of catastrophisms measured with PCS on the incidence of people with LBP for more than 3 months
Influence of fear-avoidance beliefs on 1-year incidence of chronic LBP | 1 year
  Influence of fear-avoidance beliefs measured with FABQ on the incidence of people with LBP for more than 3 months
Influence of self-efficacy on 1-year incidence of chronic LBP | 1 year
  Influence of self-efficacy measured with PSEQ-2 on the incidence of people with LBP for more than 3 months
Influence of depression on severity of LBP accroding to pain trajectories | 1 year
  Influence of depression as measured by HADS on 1 year pain trajectories recorded at the end of the study
Influence of anxiety on severity of LBP accroding to pain trajectories | 1 year
  Influence of anxiety as measured by HADS on 1 year pain trajectories recorded at the end of the study
Influence of catastrophism on severity of LBP accroding to pain trajectories | 1 year
  Influence of catastrophism as measured by PCS on 1 year pain trajectories recorded at the end of the study
Influence of fear-avoidance beliefs on severity of LBP accroding to pain trajectories | 1 year
  Influence of fear-avoidance beliefs as measured with FABQ on 1 year pain trajectories recorded at the end of the study
Influence of self-efficacy on severity of LBP accroding to pain trajectories | 1 year
  Influence of self-efficacy as measured with PSEQ-2 on 1 year pain trajectories recorded at the end of the study
Influence of depression on severity of LBP assessed with a multiaxial tool | 1 year
  Influence of depression as measured by HADS on severity as assessed with COMI, multi-axial PRO specific for LBP
Influence of anxiety on severity of LBP assessed with a multiaxial tool | 1 year
  Influence of anxiety as measured by HADS on severity as assessed with COMI, multi-axial PRO specific for LBP
Influence of catastrophism on severity of LBP assessed with a multiaxial tool | 1 year
  Influence of catastrophism as measured by PCS on severity as assessed with COMI, multi-axial PRO specific for LBP
Influence of fear-avoidance beliefs on severity of LBP assessed with a multiaxial tool | 1 year
  Influence of fear-avoidance beliefs as measured by FABQ on severity as assessed with COMI, multi-axial PRO specific for LBP
Influence of self-efficacy on severity of LBP assessed with a multiaxial tool | 1 year
  Influence of self-efficacy as measured by PSEQ-2 on severity as assessed with COMI, multi-axial PRO specific for LBP
Influence of depression on severity of LBP according to treatment use | 1 year
  Influence of depression as measured by HADS on the number of medical and paramedical appointements during the pain period
Influence of anxiety on severity of LBP according to treatment use | 1 year
  Influence of anxiety as measured by HADS on the number of medical and paramedical appointements during the pain period
Influence of catastrophism on severity of LBP according to treatment use | 1 year
  Influence of catastrophism as measured by PCS on the number of medical and paramedical appointements during the pain period
Influence of fear-avoidance beliefs on severity of LBP according to treatment use | 1 year
  Influence of fear-avoidance beliefs measured by FABQ on the number of medical and paramedical appointements during the pain period
Influence of self-efficacy on severity of LBP according to treatment use | 1 year
  Influence of self-efficacy measured by PSEQ-2 on the number of medical and paramedical appointements during the pain period
Impact of regular physical activity on LBP episode | 1 year
  Studing the impact of the intensity of physical activity during the previous month on the length and the intensity (COMI) of LBP episode.
Impact of regular physical activity on chronicity | 1 year
  Studing the impact of the intensity of physical activity during the previous month on the risk of chronicity (3 months of pain most of the day)

CONTACTS AND LOCATIONS:
Overall Officials: Stephane Genevay, MD, Principal Investigator — University Hospitals of Geneva
Locations (1):
- Geneva University Hospital, Geneva, Switzerland

REFERENCES:
- [Result] Verbunt JA, Smeets RJ, Wittink HM. Cause or effect? Deconditioning and chronic low back pain. Pain. 2010 Jun;149(3):428-430. doi: 10.1016/j.pain.2010.01.020. Epub 2010 Feb 12. No abstract available. PMID 20153582
- [Result] Buchbinder R, Batterham R, Elsworth G, Dionne CE, Irvin E, Osborne RH. A validity-driven approach to the understanding of the personal and societal burden of low back pain: development of a conceptual and measurement model. Arthritis Res Ther. 2011;13(5):R152. doi: 10.1186/ar3468. Epub 2011 Sep 20. PMID 21933393
- [Result] Maetzel A, Li L. The economic burden of low back pain: a review of studies published between 1996 and 2001. Best Pract Res Clin Rheumatol. 2002 Jan;16(1):23-30. doi: 10.1053/berh.2001.0204. PMID 11987929
- [Result] Choi BK, Verbeek JH, Tam WW, Jiang JY. Exercises for prevention of recurrences of low-back pain. Cochrane Database Syst Rev. 2010 Jan 20;2010(1):CD006555. doi: 10.1002/14651858.CD006555.pub2. PMID 20091596
- [Result] Hoy D, Bain C, Williams G, March L, Brooks P, Blyth F, Woolf A, Vos T, Buchbinder R. A systematic review of the global prevalence of low back pain. Arthritis Rheum. 2012 Jun;64(6):2028-37. doi: 10.1002/art.34347. Epub 2012 Jan 9. PMID 22231424
- [Result] Bohannon RW, Crouch R. Minimal clinically important difference for change in 6-minute walk test distance of adults with pathology: a systematic review. J Eval Clin Pract. 2017 Apr;23(2):377-381. doi: 10.1111/jep.12629. Epub 2016 Sep 4. PMID 27592691
- [Result] Kongsted A, Hestbaek L, Kent P. How can latent trajectories of back pain be translated into defined subgroups? BMC Musculoskelet Disord. 2017 Jul 3;18(1):285. doi: 10.1186/s12891-017-1644-8. PMID 28673341
- [Result] Genevay S, Marty M, Courvoisier DS, Foltz V, Mahieu G, Demoulin C, Fontana AG, Norberg M, de Goumoens P, Cedraschi C, Rozenberg S; Section Rachisde la Societe Francaise de Rhumatologie. Validity of the French version of the Core Outcome Measures Index for low back pain patients: a prospective cohort study. Eur Spine J. 2014 Oct;23(10):2097-104. doi: 10.1007/s00586-014-3325-8. Epub 2014 Jul 15. PMID 25022859
- [Result] Dionne CE, Dunn KM, Croft PR, Nachemson AL, Buchbinder R, Walker BF, Wyatt M, Cassidy JD, Rossignol M, Leboeuf-Yde C, Hartvigsen J, Leino-Arjas P, Latza U, Reis S, Gil Del Real MT, Kovacs FM, Oberg B, Cedraschi C, Bouter LM, Koes BW, Picavet HS, van Tulder MW, Burton K, Foster NE, Macfarlane GJ, Thomas E, Underwood M, Waddell G, Shekelle P, Volinn E, Von Korff M. A consensus approach toward the standardization of back pain definitions for use in prevalence studies. Spine (Phila Pa 1976). 2008 Jan 1;33(1):95-103. doi: 10.1097/BRS.0b013e31815e7f94. PMID 18165754